CLINICAL TRIAL: NCT00459472
Title: Operating Room Outcomes After Resident Training on a Virtual Reality Simulator
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left institution.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AAAA9177
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Gall Bladder Disease
Keywords: resident training; laparoscopy; virtual reality; surgical education
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Training (Other): laparoscopic training curriculum: all general surgery interns and PGY-2-5's already participate in a surgery training curriculum that includes lectures, surgery, laparoscopic training, attending surgeons evaluating performance of residents at the end of surgical procedures, written tests, and skills tests.
  Interventions: Behavioral: laparoscopic training curriculum

INTERVENTIONS:
Behavioral: laparoscopic training curriculum — All general surgery interns and PGY-2-5's already participate in a surgery training curriculum that includes lectures, surgery, laparoscopic training, attending surgeons evaluating performance of residents at the end of surgical procedures, written tests, and skills tests.

SUMMARY:
The purpose of this study is to compare outcomes of patients undergoing laparoscopic cholecystectomy before and after a laparoscopic training curriculum was implemented.

DETAILED DESCRIPTION:
All general surgery interns and PGY-2's AND PGY 3's will be enrolled in a laparoscopic surgery training curriculum that includes practicing surgical skills on a laparoscopic simulator. The PI has constructed an examination on the simulator that will document a significant level of laparoscopic skill. Each general surgery intern, second, AND THIRD year general surgery resident will be required to pass this examination on the simulator prior to being given more responsibility during cases of laparoscopic cholecystectomy. Specifically, interns, second, AND THIRD year residents must pass the examination on the simulator before they are allowed to function as primary surgeon in a supervised setting during laparoscopic cholecystectomy. These interns, PGY-2's, AND PGY 3'S would then be allowed to function as primary surgeon under the supervision of an attending surgery for laparoscopic cholecystectomy cases. The outcomes of these cases would be compared to a matched group of laparoscopic cholecystectomy cases performed by second year general surgery residents in the same supervised environment (but without having trained on the simulator) one year prior.

ELIGIBILITY:
Inclusion Criteria:

* General Surgery residents at NewYork Hospital/Columbia in PGY 1, 2, or 3.

Exclusion Criteria:

* persons who are not General Surgery residents at NewYork Hospital/Columbia in PGY 1, 2, or 3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Operative time | 1 year
Prevalence of complications (such as bile duct injuries, bilomas, infections, bleeding) | 1 year
Mortality rate | 30 days

SECONDARY OUTCOMES:
Average days of hospital stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Fowler, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States